CLINICAL TRIAL: NCT06496646
Title: Antidepressant Medication Adherence in Adults With Depression
Brief Title: Antidepressant Adherence for Depressed Adults in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 1R01MH135011-01A1 (NIH)
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Depression
Keywords: Medication adherence
MeSH Terms: conditions — Depression; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Behavioral: Arm 1 intervention
- Arm 2 (Experimental)
  Interventions: Behavioral: Arm 1 intervention; Behavioral: Arm 2 Intervention
- Arm 3 (No Intervention)

INTERVENTIONS:
Behavioral: Arm 1 intervention — This description is blinded.
  Arms: Arm 1; Arm 2
Behavioral: Arm 2 Intervention — This description is blinded
  Arms: Arm 2

SUMMARY:
The goal of this study is to test ways to help people improve their health and manage their medication for depression. This study will measure both medication adherence and depression outcomes.

DETAILED DESCRIPTION:
Participants in the study will be given a special pill bottle for depression medication. This pill bottle will track how often the bottle is opened to take medication and it will transmit that information to the research team. Participation will last 12 weeks, and will include an initial assessments over the phone and follow-up assessments over the phone or electronically approximately 6 weeks and 12 weeks later. During these assessments, a research coordinator will ask questions about your mood, quality of life, participation in the management of depression, and related topics.

ELIGIBILITY:
Inclusion Criteria:

* Penn Medicine primary care outpatients
* Clinical diagnosis of major depressive disorder
* A score of 10+ on the Patient Health Questionnaire 9 (PHQ-9)
* Age 21 to 64 years at the time of study entry
* Prescribed an antidepressant by their primary care clinician
* Express interest in taking antidepressant medication
* Own a cell phone
* Capable of using the electronic pill bottle
* English-speaking

Exclusion Criteria:

* Treated with antidepressants in the past 90 days
* Pregnant or breastfeeding
* An active substance use disorder other than nicotine
* A lifetime history of treatment for bipolar disorder or schizophrenia
* Hospital admission or emergency department visit for suicidal symptoms in the past year
* Lack capacity to provide informed consent
* Using antidepressant more than 10 days at baseline assessment

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 525 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Depression symptom response 12 weeks | 12 weeks from baseline
  A reduction of 50% in depression score from baseline as assessed by PHQ-9

SECONDARY OUTCOMES:
Antidepressant adherence | 6 and 12 weeks
  measurement of antidepressant adherence through electronic pill bottles
Depression symptom response 6 weeks | 6 weeks from baseline
  A reduction of 50% in depression score from baseline as assessed by PHQ-9

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, de-identified data from this study, including individual-level data and associated documentation, will be submitted to the NIMH Data Archive in compliance with NIMH policies. The data will be made available to qualified researchers upon request.